CLINICAL TRIAL: NCT05675657
Title: Ultrasound Guided Quadratus Lumborum Block Versus Erector Spinae Plane Block For Postoperative Analgesia In Patient Undergoing Abdominal Hysterectomy: A Randomized Double Blinded Study
Brief Title: Quadratus Lumborum Block vs Erector Spinae Plane Block in Abdominal Hysterectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Namik Kemal University (Other)
Responsible Party: Principal Investigator, Onur Baran, Assistant Professor, Namik Kemal University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2022.206.11.07
Record Dates: First submitted 2022-12-29; First posted 2023-01-09 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: Gynecologic Disease
Keywords: Erector Spinae Plane Block; Quadratus Lumborum Block; Analgesia; Abdominal Hysterectomy; Ultrasound Guidance
MeSH Terms: conditions — Genital Diseases, Female; Agnosia | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: The patients will be divided randomly by a computer-generated randomization table into three equal groups.
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control group (Placebo Comparator): Patients will be operated under general anesthesia.
  Interventions: Other: No Block
- Quadratus Lumborum Block Group (Active Comparator): Patients will receive ultrasound-guided quadratus lumborum block type III bilaterally with 30 ml of bupivacaine 0.25% on each side, totally 60 ml of bupivacaine 0.25% followed by general anesthesia.
  Interventions: Procedure: Quadratus Lumborum Block Type III
- Erector Spinae Plane Block Group (Active Comparator): Patients will receive ultrasound-guided erector spinae plane block bilaterally with 30 ml of bupivacaine 0.25% on each side, totally 60 ml of bupivacaine 0.25% followed by general anesthesia.
  Interventions: Procedure: Erector Spinae Plane Block

INTERVENTIONS:
Other: No Block — The patients will receive general anesthesia.
  Other Names: Control Group
  Arms: Control group
Procedure: Quadratus Lumborum Block Type III — Patients will receive ultrasound-guided quadratus lumborum block type III with 60 ml of bupivacaine 0.25% followed by general anesthesia.
  Other Names: QLB III
  Arms: Quadratus Lumborum Block Group
Procedure: Erector Spinae Plane Block — Patients will receive ultrasound-guided erector spinae plane block type III with 60 ml of bupivacaine 0.25% followed by general anesthesia.
  Other Names: ESPB
  Arms: Erector Spinae Plane Block Group

SUMMARY:
Postoperative pain following abdominal hysterectomy is a challenging concern as some patients suffer acute pain that could let to chronic pain over time following the surgery. Epidural analgesia which is the gold standard for postoperative pain management in abdominal surgeries including abdominal hysterectomy has side effects such as hypotension, hematoma, motor weakness of lower limbs, paresthesia, intrathecal placement of the epidural catheter and urinary retention that could prolong hospital stay. Since high frequency ultrasound machines' usage has increased in postoperative analgesia management, ultrasound guided fascial plane blocks has been performed by clinicians with high success rate. To avoid possible complications of epidural catheter placement and epidural analgesia, various techniques has been applying for an analgesic effect close to the effectiveness of epidural analgesia. These techniques include transversus abdominis plane block, rectus sheath block, wound infiltration of local anesthetics, erector spinae plane block and quadratus lumborum plane block. However, each of the plane blocks has limitations individually which prevent them to be the unique analgesic technique for postoperative analgesia following abdominal surgery. As far as the authors knowledge, there's no reported study which compares ultrasound guided erector spinae plane block versus ultrasound guided quadratus lumborum type III block (anterior quadratus lumborum block) as a preemptive analgesia technique in patients undergoing abdominal hysterectomy.

DETAILED DESCRIPTION:
Hysterectomy is one of the most frequently performed surgical procedures in the United States. The management of postoperative pain in gynecologic surgery is challenging.

Due to side effects of opioids such as nausea and vomiting, titration of opioid dosage for postoperative pain is difficult and effective postoperative analgesic regimes is needed. Ultrasound guided regional anesthesia techniques such as erector spinae plane block and quadratus lumborum block for postoperative pain management has an acceleration in usage as ultrasound guidance makes the interventions safer and easier to perform, and they contribute to better pain control and pain experience. Ultrasound guided quadratus lumborum block for postoperative pain management after abdominal surgery was firstly conceived by Blanco in 26th European Society of Regional Anesthesia Congress in 2007 as a variant of transversus abdominis plane (TAP) block. Later on he reported posterior quadratus lumborum block (QLB) in 2013 which is known as QLB II. Børglum et. al described the transmuscular quadratus lumborum block (TQL or QLB III) in 2013 which is frequently performed in abdominal wall surgeries. QLB III, transmuscular quadratus lumborum block (TQL) and anterior quadratus lumborum block; these are all synonyms and refers to injection of local anesthetic into the anterior thoracolumbar fascia (TLF) which lays between quadratus lumborum muscle and psoas major muscle. Erector spinae plane block has being performed by clinicians for abdominal and thoracic surgeries since it was firstly described by Forero et al. in 2016 for analgesia in thoracic neuropathic pain. In this ultrasound guided technique local anesthetic is applied between the transverse process of the relevant thoracic or lumbar vertebrae and the erector spinae muscle which leads to the spread of the local anesthetic cephalad, caudally and through the paravertebral space. The investigators hypothesize that performing ultrasound-guided quadratus lumborum block will be more superior or equal to erector spinae plane block in providing postoperative analgesia for patients undergoing abdominal hysterectomy under general anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* Patients who accepted to participate and signed written consent
* Aged between 18 and 75
* American Society of Anesthesiologists (ASA) physical score I or II
* Elective abdominal hysterectomy operation

Exclusion Criteria:

* Patients who declined to participate
* BMI > 35 kg/m2
* Uncontrolled systemic disease
* <18 age and >75 age
* Unable to cooperate (mental retardation)
* Low cardiac capacity
* Hypersensitivity history to the agents to be used
* Coagulopathy
* Local infections
* Opioid addiction history

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Participant eligibility is based on self-representation of gender identity who will undergo abdominal hysterectomy operation.
Enrollment: 81 (Actual)
Dates: Start 2023-01-15 (Actual); Primary Completion 2023-07-15 (Actual); Study Completion 2023-07-15 (Actual)

PRIMARY OUTCOMES:
Total dose of opioid consumption (tramadol) | in the first 24 hour postoperatively
  Total dose of tramadol consumption via patient controlled device

SECONDARY OUTCOMES:
Visual Analog Scale | measured at at 30 minute, 2, 6, 12, 24th hour postoperatively
  On a scale of 0-10, the patient will learn to quantify postoperative pain where 0= No pain and 10= Maximum worst pain.
The 1st time to rescue analgesic need | recorded within the first 24 hour postoperatively
  The time to ask for postoperative analgesia is the time from the end of operation to patient reporting Visual Analog Scale ≥ 4.
Postoperative nausea and vomiting | recorded within the first 24 hour postoperatively
  Postoperative nausea and vomiting presence

CONTACTS AND LOCATIONS:
Overall Officials: Onur Baran, Asst. Prof., Study Chair — Namik Kemal University; Ayhan Şahin, Asst. Prof., Principal Investigator — Namik Kemal University; Cavidan Arar, Prof., Study Director — Namik Kemal University
Locations (1):
- Tekirdag Namik Kemal University, Tekirdağ, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Committee Opinion No 701: Choosing the Route of Hysterectomy for Benign Disease. Obstet Gynecol. 2017 Jun;129(6):e155-e159. doi: 10.1097/AOG.0000000000002112. PMID 28538495
- [Result] Dewinter G, Teunkens A, Vermeulen K, Devroe S, Van Hemelrijck J, Meuleman C, Vergote I, Fieuws S, Van de Velde M, Rex S. Alizapride and ondansetron for the prevention of postoperative nausea and vomiting in patients undergoing laparoscopic gynaecological surgery: A double-blind, randomised, placebo-controlled noninferiority study. Eur J Anaesthesiol. 2016 Feb;33(2):96-103. doi: 10.1097/EJA.0000000000000288. PMID 26086285
- [Result] Ishio J, Komasawa N, Kido H, Minami T. Evaluation of ultrasound-guided posterior quadratus lumborum block for postoperative analgesia after laparoscopic gynecologic surgery. J Clin Anesth. 2017 Sep;41:1-4. doi: 10.1016/j.jclinane.2017.05.015. Epub 2017 Jun 1. PMID 28802593
- [Result] Sjovall S, Kokki M, Kokki H. Laparoscopic surgery: a narrative review of pharmacotherapy in pain management. Drugs. 2015 Nov;75(16):1867-89. doi: 10.1007/s40265-015-0482-y. PMID 26493289
- [Result] Sousa AM, Rosado GM, Neto Jde S, Guimaraes GM, Ashmawi HA. Magnesium sulfate improves postoperative analgesia in laparoscopic gynecologic surgeries: a double-blind randomized controlled trial. J Clin Anesth. 2016 Nov;34:379-84. doi: 10.1016/j.jclinane.2016.05.006. Epub 2016 Jun 5. PMID 27687417
- [Result] Macias AA, Finneran JJ. Regional Anesthesia Techniques for Pain Management for Laparoscopic Surgery: a Review of the Current Literature. Curr Pain Headache Rep. 2022 Jan;26(1):33-42. doi: 10.1007/s11916-022-01000-6. Epub 2022 Jan 27. PMID 35084655
- [Result] Blanco R, Ansari T, Girgis E. Quadratus lumborum block for postoperative pain after caesarean section: A randomised controlled trial. Eur J Anaesthesiol. 2015 Nov;32(11):812-8. doi: 10.1097/EJA.0000000000000299. PMID 26225500
- [Result] Gopal TVS. Ultrasound-guided transmuscular quadratus lumborum plane catheters: In the plane or out of it? Indian J Anaesth. 2019 Aug;63(8):609-610. doi: 10.4103/ija.IJA_585_19. No abstract available. PMID 31462804
- [Result] Forero M, Adhikary SD, Lopez H, Tsui C, Chin KJ. The Erector Spinae Plane Block: A Novel Analgesic Technique in Thoracic Neuropathic Pain. Reg Anesth Pain Med. 2016 Sep-Oct;41(5):621-7. doi: 10.1097/AAP.0000000000000451. PMID 27501016
- [Result] Aksu C, Sen MC, Akay MA, Baydemir C, Gurkan Y. Erector Spinae Plane Block vs Quadratus Lumborum Block for pediatric lower abdominal surgery: A double blinded, prospective, and randomized trial. J Clin Anesth. 2019 Nov;57:24-28. doi: 10.1016/j.jclinane.2019.03.006. Epub 2019 Mar 6. PMID 30851499
- [Result] Tsui BCH, Fonseca A, Munshey F, McFadyen G, Caruso TJ. The erector spinae plane (ESP) block: A pooled review of 242 cases. J Clin Anesth. 2019 Mar;53:29-34. doi: 10.1016/j.jclinane.2018.09.036. Epub 2018 Oct 3. PMID 30292068
- [Result] Chin KJ, Adhikary S, Sarwani N, Forero M. The analgesic efficacy of pre-operative bilateral erector spinae plane (ESP) blocks in patients having ventral hernia repair. Anaesthesia. 2017 Apr;72(4):452-460. doi: 10.1111/anae.13814. Epub 2017 Feb 11. PMID 28188621
- [Derived] Baran O, Sahin A, Arar C. Comparative efficacy of erector spinae plane and quadratus lumborum blocks in managing postoperative pain for total abdominal hysterectomy: A randomized controlled trial. Medicine (Baltimore). 2024 Oct 25;103(43):e40313. doi: 10.1097/MD.0000000000040313. PMID 39470511